CLINICAL TRIAL: NCT05962307
Title: Efficacy and Safety of Bulevirtide (BLV) Therapy in HDV Chronic Hepatitis (CHD) Patients in Italy: a National Real Life Data Study
Brief Title: Efficacy and Safety of Bulevirtide (BLV) Therapy in HDV Chronic Hepatitis (CHD) in Italy
Acronym: HEP4Di
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: IN-IT-589-6246
Record Dates: First submitted 2023-03-21; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-03

CONDITIONS: Hepatitis D
MeSH Terms: conditions — Hepatitis D | interventions — bulevirtide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Hepatis Delta: Bulevirtide (BLV) at a dose of 2 mg/day subcutaneously
  Interventions: Drug: Bulevirtide

INTERVENTIONS:
Drug: Bulevirtide — dose of 2 mg/day subcutaneously

SUMMARY:
Spontaneous, pharmacological observational, no-profit, retrospective, multi-center.

This study was designed to get a "real-life" snapshot across several Italian Hepatology centers. All HDV patients are followed up according to EASL 2017 guidelines. This allows uniformity on the indication for antiviral treatment and management of that antiviral therapy. No off-label medications are used. All data are retrievable from the patient's medical record. In addition, clinical and biochemical data from patients at month 0, 1, 2, 4, 6 and 12 of treatment, and otherwise within the study period, will be collected retrospectively/longitudinally.

The primary objective of the study is to describe the virological response to BLV in all patients starting BLV therapy, defined as a >2 Log decline in HDV-RNA or undetectable HDV-RNA (using the Robogene 2.0 quantitative kit, LLQ <6 IU/ml) at month 12 of therapy.

All patients with active HDV chronic hepatopathy (quantifiable HDV-RNA) who initiated treatment with BLV 2 mg/day during the study period at the S.C. Gastroenterology and Hepatology (Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico) and at participating centers, and who met the inclusion criteria and none of the exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Chronic hepatitis delta
* Compensated cirrhosis HDV related
* Bulevertide 2 mg/day within December 15, 2020, to December 31, 2022

Exclusion Criteria:

- HDV-related decompensated cirrhosis (CPT ≥7)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with active HDV chronic hepatopathy (quantifiable HDV-RNA) who initiated treatment with BLV 2 mg/day during the study period at the S.C. Gastroenterology and Hepatology (Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico) and at participating centers, and who met the inclusion criteria and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Describe the virological response to BLV in all patients starting BLV therapy | Month 12
  percentage of patients with undetectable HDV RNA.
Describe the virological response to BLV in all patients starting BLV therapy | Month 12
  percentage of patients with ≥ 2 log IU/ml decline of HDV RNA at month 12 of BLV therapy, compared to baseline.

SECONDARY OUTCOMES:
Evaluation of the percentage of patients with >2 Log decrease in HDV-RNA along with normalization of ALT, at the twelfth month of treatment | Month 12
  Percentage of patients with >2 Log decrease in HDV-RNA along with normalization of ALT
Evaluation of the percentage of patients with normal ALT, at the twelfth month of treatment | Month 12
  Percentage of patients with normal ALT at 12 months of BLV treatment
Evaluation of the percentage of patients with clinical response, i.e., the percentage of patients who remain free of liver complications, such as HCC or decompensation, at the end of the first year of treatment | Month 12
  Percentage of patients who remain free of liver complications (de novo HCC or onset of decompensation)
Evaluation of treatment safety | Month 12
  Occurrence change in serum bile acid levels (µmol/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation IRCCS Ca' Granda Ospedale Maggiore Policlinico, Division of Gastroenterology and Hepatology, Milan, Italy., Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Undecided